CLINICAL TRIAL: NCT03913000
Title: Open-label, Phase 1 Study to Investigate the Effects of Mild, Moderate, and Severe Renal Function Impairment on the Pharmacokinetics, Safety, and Tolerability of a Single Dose of ID-085
Brief Title: A Study to Evaluate ID-085 in People With Mild, Moderate, and Severe Kidney Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: ID-085-103
Record Dates: First submitted 2019-04-10; First posted 2019-04-12 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: Single-center, open-label, single-dose study is conducted in male and female subjects with renal function impairment and in healthy subjects. Groups A (mild), B (moderate), C (severe) and D (healthy subjects) will be studied in a staggered way, starting with the group with mild renal function impairment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ID-085 single dose (Experimental): Administration of the study treatment 200 mg to renally impaired subjects will be done by severity, starting with group A (mild), and followed by group B (moderate), C (severe) and D (healthy subjects).
  Interventions: Drug: ID-085

INTERVENTIONS:
Drug: ID-085 — Hard capsules for oral administration formulated at a strength of 200 mg

SUMMARY:
The primary objective of this study is to evaluate the pharmacokinetics (PK), tolerabilty and safety of a single dose of ID-085 in subjects with mild, moderate, and severe renal function impairment compared to healthy subjects

ELIGIBILITY:
Inclusion Criteria:

All subjects:

* Signed informed consent in a language understandable to the subject prior to any study-mandated procedure.
* Male and female subjects aged between 18 and 79 years (inclusive) at screening.
* Body mass index (BMI) of 18.0 to 34.0 kg/m2 (inclusive) at screening. Body weight of at least 50 kg.
* Women of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test on Day-1. They must consistently and correctly use (from at least first dosing, during the entire study, and for at least 30 days after last study treatment intake) a highly effective method of contraception with a failure rate of < 1% per year and must use condoms, diaphragm or cervical cap with spermicide, or be sexually abstinent. Hormonal contraceptive must be initiated at least 1 month before study treatment administration.

Renal function impairment subjects:

• At screening and on Day -1, the stage of renal function impairment will be defined by Creatinine Clearance (CLcr) by the Cockcroft-Gault (C-G) equation:

* Mild renal function impairment: CLcr 60-89 mL/min (Group A).
* Moderate renal function impairment: CLcr 30-59 mL/min (Group B).
* Severe renal function impairment: CLcr <30 mL/min (Group C).

The stage of renal impairment will need to be confirmed at Day -1 and the CLcr values on Day -1 will need to remain within ± 25% of the screening value.

Healthy subjects:

• Normal renal function confirmed by a CLcr ≥ 90 mL/min. Normal renal function will need to be confirmed at Day -1 and the CLcr value on Day -1 will need to remain within ± 25% of the screening value.

Exclusion Criteria:

All subjects:

* Pregnant or lactating women.
* Known hypersensitivity to ID-085 or treatments of the same class, or any of its excipients.
* Known hypersensitivity or allergy to natural rubber latex.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.

Renal function impairment subjects:

* Subjects on dialysis.
* Hemoglobin concentration < 9 g/dL.
* Serum potassium concentration > 6 mmol/L.
* Platelet count < 100 × 10^6/mL.
* History of severe renal stenosis.
* History of clinically relevant bleeding disorder.
* Gastrointestinal bleeding within 2 weeks prior to screening.
* Presence of unstable diabetes mellitus.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-08-22 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) from time zero to time t of the last measured concentration above the limit of quantification (AUC0-t) | Up to Day 3 after treatment administration
  Will be derived by non-compartmental analysis of the plasma concentration-time profiles
The plasma AUC from zero to infinity (AUC0-inf), calculated with the apparent λz | Up to Day 3 after treatment administration
  Will be derived by non-compartmental analysis of the plasma concentration-time profiles
The maximum plasma concentration (Cmax) | Up to Day 3 after treatment administration
  Will be derived by non-compartmental analysis of the plasma concentration-time profiles
The time to reach Cmax (tmax) | Up to Day 3 after treatment administration
  Will be derived by non-compartmental analysis of the plasma concentration-time profiles
Apparent total body clearance (CL/F) | Up to Day 3 after treatment administration
  Will be derived by non-compartmental analysis of the plasma concentration-time profiles
Apparent volume of distribution (Vz/F) | Up to Day 3 after treatment administration
  Will be derived by non-compartmental analysis of the plasma concentration-time profiles

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- CRS Clinical Research Services Kiel GmbH, Kiel, Germany